CLINICAL TRIAL: NCT07210775
Title: Topical Imiquimod for the Treatment of Oral Dysplastic Lesions With Clinical and Histologic Assessments
Brief Title: Topical Imiquimod Treatment of Oral Dysplasia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Anette Vistoso Monreal, Director of OralCare PreCancer and Pain Clinic, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-24-00015
Record Dates: First submitted 2025-09-18; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Oral Dysplasia; Leukoplakia Oral; Leukoplakia
Keywords: oral dysplasia; leukoplakia; prevent cancer; topical application
MeSH Terms: conditions — Leukokeratosis, Hereditary Mucosal; Leukoplakia | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients have topical imiquimod applied to oral dysplasia site (Experimental)
  Interventions: Drug: Imiquimod (topical use)

INTERVENTIONS:
Drug: Imiquimod (topical use) — Participants will be prescribed imiquimod 5% cream, with instructions to apply the cream with soft tray or gauze daily for one hour, five days a week (Monday to Friday). 6 week as one course and additional course may be added based on participant's conditions and consent. 2 follow up biopsies are scheduled 6 months and 12 months after the start of the treatment course.

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of imiquimod in treating oral dysplasia in adult patients. Imiquimod 5% cream could be a safe and practical treatment for oral epithelial dysplasia (a precancerous change in the mouth). The main questions it aims to answer are:

1. Does imiquimod help to make the lesions smaller and make the abnormal cell changes less severe?
2. How can we make this treatment safer and more feasible?

Participants will apply topical imiquimod cream to treat the oral dysplasia and receive two follow-up biopsies after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a biopsy-proven diagnosis of oral epithelial dysplasia.
* The patient is ineligible for or unwilling to undergo surgical or laser therapy.
* The patient is over 18 years old.
* The patient agrees to join the study and completes the informed consent process.

Exclusion Criteria:

* The patient has OL, and excisional surgical removal is indicated.
* The patient is immunocompromised.
* The patient is under 18 years old.
* The patient refused to join the study or did not complete the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness by Clinical Response | 52 weeks after the start of the participant's treatment course
  Clinical response: Change in the size of the lesion. Measurement of the lesion and scored according to RECIST criteria
Effectiveness by histopathological assessment | 52 weeks after the start of participant's treatment course
  Evaluation of the changes of degree of dysplasia following the WHO three-tier grading of oral dysplasia in which Oral epithelial dysplasia is graded as mild, moderate, and severe.

SECONDARY OUTCOMES:
Frequency of Adverse Effects | 24 months
  Percentage of participants experienced at least 1 adverse events
Manageability of Adverse effects | 24 months
  Percentage of adverse effect can not be managed by OTC medication
Treatment Adherence | 24 months
  Percentage of patient with treatment adherence (≥80% Day adherence)

CONTACTS AND LOCATIONS:
Locations (1):
- OralCare PreCancer and Pain Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sroussi H, Villa A, Alhadlaq MA, Ikeda K, Veluppillai S, Treister N, Monreal AV, Vacharotayangul P, Lodolo M, Woo SB. Imiquimod for the treatment of oral leukoplakia: A two-center retrospective study. Oral Dis. 2025 Feb;31(2):444-451. doi: 10.1111/odi.15069. Epub 2024 Jul 15. PMID 39007165